CLINICAL TRIAL: NCT05203653
Title: Effectiveness of Aerobic Exercise to Mitigate Hyperglycemia After Fasted Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115197
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes
Keywords: resistance exercise, aerobic exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will undergo two separate testing sessions
  Interventions: Behavioral: Resistance exercise only; Behavioral: Resistance exercise plus cool down

INTERVENTIONS:
Behavioral: Resistance exercise only — Participants will perform 3 sets of 8 repetitions of 7 different exercises while in a fasted state.
Behavioral: Resistance exercise plus cool down — Participants will perform 3 sets of 8 repetitions of 7 different exercises while in a fasted state followed by a 10-minute light aerobic cool down

SUMMARY:
Certain types and timings of exercise are known to cause hyperglycemia (high blood glucose) in people with type 1 diabetes. Hyperglycemia increases the risk of most long-term complications for individuals with this complication. However, using insulin corrections to treat post-exercise hyperglycemia can increase the risk of late-onset hypoglycemia (low-blood glucose).

Anaerobic activities performed in a fasted state are known to cause increases in blood glucose and post-exercise hyperglycemia in most individuals with type 1 diabetes. This study proposes to examine the effect of a ten-minute aerobic cool down after resistance exercise on the blood glucose response to fasted exercise of individuals with type 1 diabetes. It is hypothesized that adding a short aerobic cool down at the end of a fasted resistance exercise session will attenuate post-exercise increases in blood glucose observed in previous studies, leading to less post-exercise hyperglycemia.

DETAILED DESCRIPTION:
Individuals with type 1 diabetes (T1D), are at elevated risk of low muscular strength, as well as accelerated decline in muscle strength and functional status with aging. Resistance exercise (RE) is a proven intervention that has been demonstrated to improve physical function, muscle mass, body composition, mental health, bone mineral density, insulin sensitivity, blood pressure, lipid profiles, and cardiovascular health for all adults. Clinical guidelines recommend that individuals with T1D perform RE twice weekly to optimally benefit from RE yet most individuals with T1D are unable to meet these recommendations. Two barriers to exercise responsible for this discrepancy are a fear of hypoglycemia from exercise, and a loss of control over diabetes. To limit barriers to exercise, much research has been done to identify exercise modalities that have minimal risk for hypoglycemia, including recent investigations demonstrating a blood glucose increase leading to hyperglycemia in response to RE while participants are fasted. Hyperglycemia frequency is directly related to the incidence of diabetes-related complications, so exercise recommendations should minimize risk of hyperglycemic and hypoglycemic responses. Clinical guidelines for post-exercise hyperglycemia recommend a corrective insulin dose or a brief aerobic cool down, however the efficacy of an aerobic cool down has yet to be empirically tested. Additionally, overcorrection of hyperglycaemia with insulin after exercise can result in an increased risk of severe late onset hypoglycaemia, which could even be fatal.

The study will have a randomized, repeated measures design with two testing sessions (one with a cool down and one without a cool down) in addition to a baseline fitness assessment. Interested participants will be invited to the Physical Activity and Diabetes Laboratory on the main campus of the University of Alberta. Participants will be asked questions related to diabetes care, physical activity levels, and medication. Blood pressure and heart rate will also be measured. Where participants are eligible, anthropometric characteristics will be measured using standard protocols. Those who meet all eligibility criteria and complete informed consent forms will be asked to complete the initial exercise tests. Participants will perform a submaximal aerobic capacity test to extrapolate the participant's aerobic capacity. Participants will also undergo a strength test for each of the seven exercises involved in the study, in order to estimate the maximum weight they can move for 3 sets of 8 repetitions (8RM). During this session the investigators will introduce participants to the activity monitor (accelerometer) that will be worn on the day before, the day of, and the day after each testing session. The accelerometer will provide information on background physical activity and sleep patterns that might act as confounders where the blood glucose responses to exercise are concerned.

Testing sessions: Participants will be asked to arrive at the lab between 7:00 and 8:00 am for both sessions, which will be randomly assigned by tossing a fair coin. During the sessions, participants will be asked to perform a total of seven resistance exercises (leg press, chest press, leg curls, lat pulldowns, seated row, shoulder press, and abdominal crunches). The protocol will be 3 sets of 8 repetitions at the participant's 8 RM. Participants will be asked to match their daily food and insulin intake as closely as possible from one testing session to the next for the day before, day of and day after the testing session. During this time participants will also wear an accelerometer on their waist during the day, and on their non-dominant wrist at night. Participants will be provided with log sheets to assist in both of these tasks and will also be asked to avoid strenuous exercise and alcohol intake.

A CGM sensor will be subcutaneously inserted by one of the investigators (trained by a group from the CGM manufacturer) into the anterior abdominal area of the participant approximately 2 days prior to the first testing session. The Dexcom G6 CGM will store glucose data every 5 minutes for up to 10 days. The participant will be instructed on how to remove their sensor at least 24 hours after the exercise session, and will be asked to upload their data to Dexcom Clarity to share with the study team. If the participant habitually uses their Dexcom G6 in their diabetes care, they will be provided with the option to start their own CGM for the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 diabetes for more than 12 months
* using either multiple daily insulin injections or continuous subcutaneous insulin infusion
* willing and able to perform resistance exercise
* HbA1c < 10.0%
* ability to attend laboratory-based sessions at the University of Alberta in Edmonton

Exclusion Criteria:

* HbA1c >9.9%
* Frequent and unpredictable hypoglycaemia
* A change in insulin management strategy within two months of the study
* blood pressure > 144/95
* severe peripheral neuropathy
* a history of cardiovascular disease
* musculoskeletal injuries affecting the ability to perform resistance exercise.
* treatment with medications (other than insulin) that affect glucose metabolism (e.g. atypical antipsychotics, corticosteroids)
* body mass index >30kg/m2
* smoking
* moderate to high alcohol intake (>2 drinks per day)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
percent time spent in hyperglycemia | 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  amount of time spent with interstitial glucose (measured by continuous glucose monitoring) greater than 9.9 mmol/L

SECONDARY OUTCOMES:
mean continuous glucose monitoring (CGM) glucose | 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  mean values of interstitial glucose levels measured by CGM
frequency of hyperglycemia | 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  number of times that CGM glucose is equal to or greater than 10.0 mmol/L
frequency of hypoglycemia | 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  number of times that CGM glucose is equal to or lower than 3.9 mmol/L
percent time spent in hypoglycemia | 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  percentage of time that CGM glucose is equal to or less than 3.9 mmol/L
percent time in range | 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  percentage of time that CGM glucose is between 4.0 and 9.9 mmol/L
capillary glucose | from 0 minutes to 45 minutes (during exercise)
  change in capillary glucose during exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No